CLINICAL TRIAL: NCT03812393
Title: Phase II Trial Evaluating the Efficacy and Safety of Neoadjuvant Neratinib and Chemotherapy in Early Stage Triple-Negative Breast Cancer Patients Who Exhibit Enhanced HER2 Signaling by Live Cell HER2 Signaling Transduction Analysis (FACT-2)
Brief Title: Evaluating the Efficacy of Neratinib on Live Cell HER2 Signaling Transduction Analysis Positive Triple Negative Breast
Acronym: FACT-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: West Cancer Center (Other)
Collaborators: Celcuity Inc (Industry); Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002
Record Dates: First submitted 2019-01-08; First posted 2019-01-23 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Triple Negative Breast Cancer; Early-stage Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — neratinib

STUDY DESIGN:
Intervention Model Description: single-arm interventional clinical trial with an early check for futility using a surrogate endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): TNBC patients with HER2 signal positive are treated with neratinib for 3 weeks followed by 12 weeks of neratinib in combination with weekly paclitaxel and carboplatin
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — For cycle 1 subjects will receive Neratinib 240mg daily for 21 days. For cycle 2-5, subjects will receive carboplatin AUC of 1.5 and Paclitaxel 80mg/m2 on day one in combination with Neratinib 240mg daily for 21 day.
  Other Names: Live Cell HER2 signaling Transduction Analysis (CELx)

SUMMARY:
An Open-Label Phase II Trial to Evaluate the Efficacy and Safety of Neoadjuvant Neratinib Followed by Weekly Paclitaxel and Carboplatin Plus Neratinib in Early Stage Triple-Negative Breast Cancer Patients Who Exhibit Enhanced HER2 Signaling by Live Cell HER2 Signaling Transduction Analysis (FACT-2)

DETAILED DESCRIPTION:
This is a prospective, single arm, open label, interventional study designed to evaluate the efficacy of neoadjuvant chemotherapy with a pan-HER inhibitor in patients with ER-/PR-/HER2-(triple-negative) invasive breast cancer who have abnormal HER2-driven signaling activity determined by the Celcuity CELx HER2 signal function (HSF) test. Patients will be required to have a prescreening research core needle biopsy to procure a fresh tumor specimen that will be sent to Celcuity for CELx HSF testing, in order to assess the status of their HER2-driven signaling activity (abnormally or normally active). While waiting for results of the CELx HSF test, patients may receive the first dose of weekly paclitaxel at the investigator's discretion. Patients whose CELx HSF test indicate they have abnormal HER2-driven signaling activity will then receive neratinib as a single agent daily for 21 days and then neratinib plus paclitaxel and carboplatin.

The primary endpoint of the study is to evaluate whether patients with triple-negative breast cancers (estrogen (ER) and progesterone (PR) receptors < 10%; HER2-negative per standard ASCO/CAP testing criteria), but with abnormal HER2-driven signaling pathways determined by the Celcuity CELx HSF assay, and who receive HER2-targeted therapy with neoadjuvant chemotherapy will have a higher rate of pathological complete response (pCR) in the breast and lymph nodes (pCR breast and lymph nodes) than has been found historically in patients with triple-negative breast cancer who have received neoadjuvant chemotherapy. Secondary endpoints include pathologic complete response (breast), clinical complete response (cCR), residual cancer burden (RCB) 0-1 index, and relationship between quantitative CELx score and pCR rate.

It is expected that approximately 135 patients will need to be prescreened in order to enroll 27 patients who have abnormal HER2-driven signaling activity.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and must have signed and dated an appropriate IRB-approved consent form that conforms to federal and i institutional guidelines for the pre-entry research core biopsy for CELx HSF testing and for initiating chemotherapy
* Patients must be female.
* Patients must be ≥ 18 years old.
* Patient must have an ECOG performance status of 0 or 1
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy.
* The primary breast tumor must be palpable and measure ≥ 1.0 cm on physical exam.
* The regional lymph nodes can be cN0 or cN1
* The tumor size can be T1c or T2
* Ipsilateral axillary lymph nodes must be evaluated by imaging (mammogram, ultrasound, and/or MRI) within 6 weeks prior to initiating chemotherapy. If suspicious or abnormal, FNA or core biopsy is recommended, also within 6 weeks prior to initiating chemotherapy. Findings of these evaluations will be used to determine the nodal status prior to initiating chemotherapy.

  * Nodal status - negative

    * Imaging of the axilla is negative;
    * Imaging is suspicious or abnormal but the FNA or core biopsy of the questionable node(s) on imaging is negative;
  * Nodal status - positive

    * FNA or core biopsy of the node(s) is cytologically or histologically suspicious or positive.
    * Imaging is suspicious or abnormal but FNA or core biopsy was not performed.
* Tumor specimen obtained at the time of diagnosis must have estrogen (ER) and progesterone (PR) receptors < 10%.
* Tumor specimen obtained at the time of diagnosis must have been determined to be HER2-negative as follows:

  * Immunohistochemistry (IHC) 0-1+; or
  * IHC 2+ and ISH non-amplified with a ratio of HER2 to CEP17 < 2.0, and if reported, average HER2 gene copy number < 4 signals/cells; or
  * ISH non-amplified with a ratio of HER2 to CEP17 < 2.0, and if reported, average HER2 gene copy number < 4 signals/cells.
* Blood counts performed within 6 weeks prior to initiating chemotherapy must meet the following criteria:

  * Absolute neutrophil count (ANC) must be ≥ 1200/mm3;
  * platelet count must be ≥ 100,000/mm3; and
  * hemoglobin must be ≥ 10 g/dL.
* The following criteria for evidence of adequate hepatic function performed within 6 weeks prior to initiating chemotherapy must be met:

  * total bilirubin must be ≤ upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * alkaline phosphatase must be ≤ 2.5 x ULN for the lab; and
  * AST must be ≤ 1.5 x ULN for the lab.
  * Alkaline phosphatase and AST may not both be > the ULN. For example, if the alkaline phosphatase is > the ULN but ≤ 2.5 x ULN, the AST must be ≤ the ULN. If the AST is > the ULN but ≤ 1.5 x ULN, the alkaline phosphatase must be ≤ ULN. Note: If ALT is performed instead of AST (per institution's standard practice), the ALT value must be ≤ 1.5 x ULN; if both were performed, the AST must be ≤ 1.5 x ULN.
* Patients with AST or alkaline phosphatase > ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET-CT, or PET scan) performed within 6 weeks prior to initiating chemotherapy does not demonstrate metastatic disease and the requirements in criterion 4.2.13 are met.
* Patients with alkaline phosphatase that is > ULN but ≤ 2.5 x ULN or unexplained bone pain are eligible for inclusion in the study if a bone scan, PET-CT scan, or PET scan performed within 6 weeks prior to initiating chemotherapy does not demonstrate metastatic disease.
* Serum creatinine performed within 6 weeks prior to initiating chemotherapy must be ≤ 1.5 x ULN for the lab.
* The left ventricular ejection fraction (LVEF) assessment by echocardiogram or MUGA scan performed within 90 days prior to initiating chemotherapy must be ≥ 50% regardless of the facility's lower limit of normal (LLN).
* Patients with reproductive potential must agree to use an effective non-hormonal method of contraception during therapy, and for at least 7 months after the last dose of study therapy.
* Patients are candidates for weekly paclitaxel and carboplatin chemotherapy as determined by treating physician.
* Patients with multifocal breast cancer are included as long as none of the tumors are HER2 positive by IHC or FISH and targeted lesion meets current inclusion criteria.
* Conditions for patient eligibility (Study Enrollment) A patient cannot be considered eligible for this study unless all of the following conditions are met:
* The patient must have consented to participate and must have signed and dated an appropriate IRB-approved consent form that conforms to federal and institutional guidelines for the FACT-2 study treatment.
* Tumor determined to have abnormal HER2-driven signaling activity based on the CELx HSF test.

Exclusion Criteria:

* T3 or T4 tumors including inflammatory breast cancer.
* FNA alone to diagnose the breast cancer.
* Excisional biopsy or lumpectomy performed prior to initiating chemotherapy.
* Surgical axillary staging procedure prior to initiating chemotherapy. Pre- neoadjuvant therapy sentinel node biopsy is not permitted. (FNA or core biopsy is acceptable.)
* Definitive clinical or radiologic evidence of metastatic disease. Required imaging studies must have been performed within 6 weeks prior to initiating chemotherapy.
* Synchronous bilateral invasive breast cancer. (Patients with synchronous and/or previous contralateral DCIS or LCIS are eligible.)
* Any previous history of ipsilateral invasive breast cancer or ipsilateral DCIS. (Patients with synchronous or previous ipsilateral LCIS are eligible.)
* Previous therapy with anthracycline, taxanes, trastuzumab, or other HER2 targeted therapies for any malignancy.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy, etc. (These patients are eligible if this therapy is discontinued prior to initiating chemotherapy.)
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 2 years prior to initiating chemotherapy.
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens. This includes but is not confined to:

  * Active cardiac disease:

    * angina pectoris that requires the use of anti-anginal medication;
    * ventricular arrhythmias except for benign premature ventricular contractions;
    * supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication;
    * conduction abnormality requiring a pacemaker;
    * valvular disease with documented compromise in cardiac function; and
    * symptomatic pericarditis.
  * History of cardiac disease:

    * myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function;
    * history of documented congestive heart failure (CHF); and
    * documented cardiomyopathy.
* Uncontrolled hypertension defined as sustained systolic BP > 150 mmHg or diastolic BP > 90 mmHg. (Patients with initial BP elevations are eligible prior to initiating chemotherapy if initiation or adjustment of BP medication lowers pressure.)
* Active hepatitis B or hepatitis C with abnormal liver function tests.
* Intrinsic lung disease resulting in dyspnea.
* Poorly controlled diabetes mellitus.
* Active infection or chronic infection requiring chronic suppressive antibiotics.
* Patients known to be HIV positive.
* Nervous system disorder (paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) ≥ grade 2, per the CTCAE v4.0.
* Malabsorption syndrome, ulcerative colitis, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal function.
* Other non-malignant systemic disease that would preclude treatment with any of the treatment regimens or would prevent required follow-up.
* Conditions that would prohibit administration of corticosteroids.
* Chronic daily treatment with corticosteroids with a dose of ≥ 10 mg/day methylprednisolone equivalent (excluding inhaled steroids).
* Known hypersensitivity to any of the study drugs or any of the ingredients or excipients of these drugs (e.g., Cremophor® EL), including sensitivity to benzyl alcohol.
* Pregnancy or lactation at the initiation of chemotherapy. (Note: Pregnancy testing must be performed within 2 weeks prior to initiating chemotherapy according to institutional standards for women of childbearing potential).
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Evidence after a clinical examination that the subject's tumor is progressing after treatment with one week of paclitaxel and before a CELx HSF test result is available.
* For participation in adherence monitoring: no access to the web via smart phone, tablet or computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients experiencing ≥ 20% response to neratinib only therapy | 4 weeks
  patient with HER2 positive signal by CELx will be exposed to neratinib to determine response to HER2 therapy
rate of pathologic complete response (pCR) | 15 weeks
  percentage of patients with no tumor in breast at surgery following study treatment

SECONDARY OUTCOMES:
Clinical complete response (cCR) | 15 weeks
  Endpoint Definition: Percentage of patients with clinical complete response rate based on physical examination of the breast and axilla.
Residual cancer burden (RCB) 0-1 | 15 weeks
  The measure of the amount of tumor left in breast at surgery following study treatment
The PCR rate in patients experiencing greater than or equal to 20% reduction in tumor volume following treatment with neratinib only in cycle 1. | 15 weeks
  To determine whether a significant decrease in size of tumor can predict whether the rate of complete tumor killing at surgery following study treatment
Safety and Toxicity per NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0). | 15 weeks
  Measure whether the study treatment is safe and tolerable
Increase in the number of patients completing neratinib prescription with the use of web based symptom monitoring | 15 weeks
  See whether mobile application that connects patient at home to treatment team could increase patients ability to complete drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Vidal, MD.,PhD, Principal Investigator — West Cancer Center
Locations (1):
- West Cancer Center, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang Y, Burns DJ, Rich BE, MacNeil IA, Dandapat A, Soltani SM, Myhre S, Sullivan BF, Furcht LT, Lange CA, Hurvitz SA, Laing LG. A functional signal profiling test for identifying a subset of HER2-negative breast cancers with abnormally amplified HER2 signaling activity. Oncotarget. 2016 Nov 29;7(48):78577-78590. doi: 10.18632/oncotarget.12480. PMID 27713176
- [Result] Huang Y, Burns DJ, Rich BE, MacNeil IA, Dandapat A, Soltani SM, Myhre S, Sullivan BF, Lange CA, Furcht LT, Laing LG. Development of a test that measures real-time HER2 signaling function in live breast cancer cell lines and primary cells. BMC Cancer. 2017 Mar 16;17(1):199. doi: 10.1186/s12885-017-3181-0. PMID 28302091